CLINICAL TRIAL: NCT05789433
Title: Effects of Aerobic Exercise on Skeletal Muscle Remodeling in Colorectal Cancer
Acronym: RESTORE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: AdventHealth Translational Research Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Justin Brown, Director, Exercise & Cancer Biology Research Program, AdventHealth Translational Research Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: PBRC 2022-014; R01CA270274 (NIH)
Record Dates: First submitted 2023-03-16; First posted 2023-03-29 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Colonic Neoplasms; Rectal Neoplasms
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Attention control (Sham Comparator): Static stretching
  Interventions: Behavioral: Progressive stretching
- Aerobic exercise (Experimental): Aerobic exercise at a dose of 225 minutes per week
  Interventions: Behavioral: Aerobic exercise

INTERVENTIONS:
Behavioral: Aerobic exercise — Moderate- to vigorous-intensity aerobic exercise
  Arms: Aerobic exercise
Behavioral: Progressive stretching — Statistic stretching of eight major muscle groups
  Arms: Attention control

SUMMARY:
The goal of this clinical trial is to quantify the effects of aerobic exercise training compared to attention control on intermuscular adipose tissue in colorectal cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Histologically confirmed stage I, II, or III colon or rectal cancer
* Completed surgical resection with curative intent
* Completed other cancer-directed treatments
* Engage in <150 minutes per week of moderate- to vigorous-intensity structured endurance exercise
* No planned major surgery during the study period
* Readiness to exercise, as determined by a modified version of the Physical Activity Readiness Questionnaire
* Ability to provide written informed consent
* Provide written approval by a qualified healthcare professional
* Willing to be randomized

Exclusion Criteria:

* Evidence of metastatic or recurrent colorectal cancer
* Concurrently actively treated other (non-colorectal) cancer
* Scheduled to receive other postoperative cancer-directed treatment(s)
* Currently pregnant, breastfeeding, or planning to become pregnant within the next 24 weeks
* Currently participating in another study with competing outcomes
* Contraindications to magnetic resonance imaging
* Any dietary condition or restriction that would limit tolerance of a mixed meal challenge
* Any other cardiovascular, pulmonary, orthopedic, neurologic, psychiatric, or other condition that, in the investigator's opinion, would preclude participation or successful compliance with the protocol
* Any other situation that, in the opinion of the investigator, would negatively impact subject safety or successful compliance with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Whole-Body Intermuscular Adipose Tissue | up to Week 12
  Mean (kg) whole-body intermuscular adipose tissue quantified using magnetic resonance imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Justin C. Brown, Ph.D., Principal Investigator — AdventHealth
Locations (1):
- AdventHealth, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes